CLINICAL TRIAL: NCT07095049
Title: A Phase1, Randomized, Double-Blind, Placebo-Controlled Study of Single, Twice Daily (BID), and Repeated Dosing of Ascending Doses, to Evaluate Safety, Tolerability, and Systemic Exposure of Intranasal Administration Apo-Si-K170A-C76 in Healthy Subjects.
Brief Title: Safety, Tolerability, and Systemic Exposure of Apo-Si- K170A-C76 in Healthy Volunteers
Acronym: BID
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Interna Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sir-001
Record Dates: First submitted 2025-06-22; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: SARS-CoV-2 (COVID-19) Infection
Keywords: SARS-CoV-2; First in Human; Safety; Tolerability; Systemic Exposure
MeSH Terms: conditions — COVID-19; Infections | interventions — C 76; Polychlorinated Biphenyls

STUDY DESIGN:
Intervention Model Description: The study is composed of 7 dosing cohorts. Cohorts #1-3 for single ascending doses; Cohorts #4-5 for BID ascending doses; Cohorts #6-7 for repeated BID dosing for 5 consecutive days, of ascending doses.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal Apo-Si-K170A-C76 Solution of 20 mg/ml in 5% glucose, 0.5% Benzyl Alcohol (BA) in water (Experimental): Intervention drug intranasal administration
  Interventions: Drug: Apo-Si-K170A-C76
- 5% glucose, 0.5% benzyl alcohol in RNase free water (Placebo Comparator): Intranasal
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apo-Si-K170A-C76 — Apo-Si-K170A-C76 is an small interfering RNA (siRNA) against SARS-CoV-2
  Other Names: c76
  Arms: Intranasal Apo-Si-K170A-C76 Solution of 20 mg/ml in 5% glucose, 0.5% Benzyl Alcohol (BA) in water
Drug: Placebo — 5% glucose, 0.5% benzyl alcohol in RNase free water
  Other Names: pcb
  Arms: 5% glucose, 0.5% benzyl alcohol in RNase free water

SUMMARY:
The goal of this First in Human Phase 1 clinical trial is to to assess the safety, tolerability, and systemic exposure of single, twice daily (BID) doses and repeated BID doses of ascending dosing by intranasal administration of Apo-Si-K170AC76 in healthy adult subjects. The primary objective is to evaluate the safety and tolerability of single, BID, and repeated BID, ascending dosing of Apo-Si-K170A-C76 administered intranasally (IN) in healthy adult subjects.

The secondary objective is to evaluate the systemic exposure to Apo-Si-K170A-C76 following intranasal administration in healthy adult subjects under the aforementioned administration regimens. Researchers will compare the active drug Apo-Si-K170A-C76 to placebo control.

DETAILED DESCRIPTION:
Upon signing the informed consent, the subjects underwent a screening period for eligibility evaluation. Subjects were admitted to the Research Unit on Day 1 and eligibility was confirmed again. Eligible subjects, as determined by the Principal Investigator (PI), were randomized as close as possible prior to1st drug administration on Day 1, to receive either intranasal Apo-Si-K170A-C76 or matching placebo. Dosing depended on the cohort the subjects were assigned to.

Intranasal (IN) administration was performed to both nostrils of all participants.

The nasal spray device contains the Study Drug at 20 mg/mL and delivers 0.1 mL volume per actuation. The subjects received 1-3 actuations per nostril alternately, according to dosing group. Thus, during each administration cohort, dosages registered as dose/nostril are received twice per subject, one dose to each nostril.

The study was composed of 7 dosing cohorts. Administration in cohorts 1-5 took place on Day 1. Administration to cohorts 6-7 took place from Day 1 to Day 5. The study drug (or placebo) was administered to both nostrils via intranasal spray, while the subject is seated. All subjects arrived at the clinic for a follow up visit 7±2 days after last day of administration.

Cohort 1 involved an initial administration of a single (low) dose of Apo-Si-K170A-C76 (2mg/100μl/nostril, to both nostrils). Cohort 2 involved administration of a single dose of Apo- Si-K170A-C76 at a double dose of the first dose (4mg/200μl/nostril, to both nostrils). Cohort 3 involved administration of a single dose of Apo-Si-K170AC76 at the target dose (x3 of first dose, 6mg/300μl/nostril, to both nostrils).

Cohort 4 involved BID administration of the same dose as cohort 2, and cohort 5 involved BID administration of the same dose as cohort 3. All BID dosing was separated by 6 hours.

Cohort 6 involved administration of repeated BID doses of Apo-Si-K170A (at the same dose level or lower than that administered in Cohort 4) taken from Day 1 to Day 5. Cohort 7, which aims to reach target dose, involved administration of repeated BID doses of Apo-Si-K170A-C76 (at the same dose level or lower than that administered in Cohort 5) taken also from Day 1 to Day 5.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants must be ≥ 18 years old.
* Understands the study procedures described in the Informed Consent Form (ICF), be willing and able to comply with the protocol, and provides written consent.
* Not pregnant or lactating and willing to comply with the contraceptive requirements from enrolment to 3 months post last dose. Contraceptive requirements include the following:
* Use a condom with a spermicide to prevent pregnancy in a female partner or to prevent exposure of any partner (male and female) to the study intervention treatment.
* Male sterilization with the appropriate post vasectomy documentation of the absence of sperm in the ejaculate (please note that the use of condom with spermicide will still be required to prevent partner exposure). This applies only to males participating in the study.
* In addition, for female partners and female participants of childbearing potential, must use another form of contraceptive such as one of the highly effective methods (pills, Intra Uterine Device (IUD)).
* True abstinence - sexual abstinence is considered as a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments.

The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.

* In addition to the contraceptive requirements above, male subjects must agree not to donate sperm for 3 months post last dose of treatment.
* Subject is in good health with no history of clinically significant medical conditions (as described in Exclusion criteria) that would interfere with subject safety, as defined by relevant medical history, physical examination and routine laboratory tests, and ECG, and as determined by the investigator at an admission evaluation.
* Subjects will have documented relevant medical history prior to entering the study and/or following relevant medical history review with the study physician at screening.

Exclusion Criteria:

* History or evidence of any clinically significant or currently active cardiovascular, (including thromboembolic events), respiratory, dermatological, gastrointestinal, endocrine, hematological, hepatic, immunological, rheumatological, metabolic, urological, renal, neurological, or psychiatric illness. Specifically:
* Subjects with any history of physician diagnosed and/or objective test-confirmed asthma, chronic obstructive pulmonary disease, pulmonary hypertension, reactive airway disease, or chronic lung condition of any etiology or who have experienced:

  * Significant/severe wheeze in the past
  * Respiratory symptoms including wheeze which have ever resulted in hospitalization.
  * Known bronchial hyper-reactivity to viruses.
* History of thromboembolic, cardiovascular, or cerebrovascular disease
* History or evidence of diabetes mellitus
* Any concurrent serious illness, including history of malignancy that could interfere with the aims of the study or a subject completing the study. Basal cell carcinoma within 5 years of treatment or with evidence of recurrence is also an exclusion.
* Migraine with associated neurological symptoms such as hemiplegia or vision loss. Cluster headache/migraine or prophylactic treatment for migraine.
* History or evidence of autoimmune disease or known immunodeficiency of any cause.
* Other major diseases that, in the opinion of the investigator, could interfere with a subject completing the study and necessary investigations.
* Immunosuppression of any type.
* Any significant abnormality altering the anatomy or function of the nose or nasopharynx in a substantial way (including loss of or alterations in smell or taste), a clinically significant history of epistaxis (large nosebleeds) within the last 3 months, nasal or sinus surgery within 6 months pre-screening.
* Clinically active rhinitis (including hay fever) or history of moderate to severe rhinitis, or history of seasonal allergic rhinitis likely to be active at the time of inclusion into the study and/or requiring regular nasal corticosteroids on at least a weekly basis, within 30 days prior to screening.
* History of anaphylaxis and/or a history of severe allergic reaction or significant intolerance to any food or drug, as assessed by the PI.
* History or presence of alcohol addiction, or excessive use of alcohol. The subject has a history of consuming more than 7 units of alcoholic beverages per week for male subjects and more than 5 units for females (Note: one unit = 330 mL of beer, 110 mL of wine, or 28 mL of spirits), or has a history of alcoholism or drug/chemical/substance abuse within the past 2 years prior to screening.
* Psychiatric illness, including subjects with a history of depression and/or anxiety with associated severe psychiatric comorbidities, for example psychosis. Specifically, (a) Subjects with history of anxiety-related symptoms of any severity within the last 2 years if the Generalized Anxiety Disorder-7 score is ≥4; (b) Subjects with a history of depression of any severity within the last 2 years if the Patient Health Questionnaire- 9 score is ≥4
* Subjects who have smoked ≥5 pack years at any time [5 pack years is equivalent to one pack of 20 cigarettes a day for 5 years]). For subjects who have smoked <5 pack years at any time, in the 3 months prior to screening, exclusion will apply if they have used tobacco in any form (e.g. smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch) or electronic cigarettes.
* A Body Mass Index (BMI) ≤18 Kg/m2 and ≥28 Kg/m2. The upper limit of BMI may be increased up to 30 Kg/m2 at the PI's discretion, in the case of physically fit muscular individual.
* Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
* At the discretion of the PI, any clinically significant abnormal finding on screening biochemistry, hematology, serology , microbiology blood tests or urinalysis or
* Positive HIV, active/chronic hepatitis B or C test.
* Positive human chorionic gonadotropin (β-HCG) or positive alcohol test
* Confirmed positive test for drugs of abuse and/or urinary cotinine at screening and on admission (Day 1).
* Twelve-lead ECG recording with clinically relevant abnormalities as judged by the study physician/PI.
* Presence of cold-like symptoms and/or fever (defined as subject presenting with a temperature reading of >37.9ºC) at screening or on admission (Day 1).
* Receipt of blood or blood products, or loss (including blood donations) of 550 mL or more of blood during the 3 months prior to screening.

Exclusion Criteria regarding Medications:

* Use of any medication or product (prescription or over-the-counter) for symptoms of hay fever, nasal congestion or respiratory tract infections, or dermatitis/eczema including the use of regular nasal or medium-high potency dermal corticosteroids, antibiotics and First Defence™ (or generic equivalents) within 7 days prior to screening. The sporadic use of paracetamol or other medications will be acceptable only as agreed by the PI.
* Receipt of any investigational drug within 3 months prior to screening.
* Receipt of three or more investigational drugs within the previous 12 months prior to screening.
* Receipt of systemic (intravenous and/or oral) glucocorticoids or systemic antiviral drugs within 6 months prior to screening.
* Over-the-counter medications (e.g., paracetamol or ibuprofen) where the dose taken over the preceding 7 days prior to screening had exceeded the maximum permissible 24-hour dose (e.g., >4g per day of paracetamol over the preceding week).
* Chronically used medications, including any medication known to be a moderate/potent inducer or inhibitor of cytochrome P450 enzymes, within 21 days prior to screening.
* Subjects who have received any systemic chemotherapy agent, immunoglobulins, or other cytotoxic or immunosuppressive drugs at any time.

General Exclusion Criteria:

* Subjects who are currently employed by or are first-degree relative of someone employed by the Sponsor or participating clinical trial site, or any Contract Research Organization involved in this study.
* Any other reason that the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability, as evaluated by Adverse Events (AEs) classification, following single, twice-daily (BID) and repeated BID ascending doses of Apo-Si-K170A-C76 following IN in healthy participants. | 5 days
  Adverse events (AE) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, most updated version) terminology and presented in tables by System Organ Class (SOC). AE data will be listed individually and summarized by SOC and by Preferred Term (PT) within a system organ class.
The safety and tolerability, as evaluated by Treatment-Emergent Adverse Events (TEAEs) frequency, following single, twice-daily (BID) and repeated BID ascending doses of Apo-Si-K170A-C76 following IN in healthy participants. | 5 days
  Frequency of TEAEs and drug-related adverse events will be summarized in tables by SOC, PT and by seriousness.
The safety and tolerability, as evaluated by AEs classification, blood tests and other physiological parameters, following single, twice-daily (BID) and repeated BID ascending doses of Apo-Si-K170A-C76 following IN in healthy participants. | 5 days
  Adverse events (AE) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, most updated version) terminology and presented in tables by System Organ Class (SOC). AE data will be listed individually and summarized by SOC and by Preferred Term (PT) within a system organ class.
  Frequency of Treatment-Emergent Adverse Events (TEAEs) and drug-related adverse events will be summarized in tables by SOC, PT and by seriousness. Concomitant medications entered into the database will be coded using the public World Health Organization (WHO) Drug Reference List, which employs the Anatomical Therapeutic Chemical classification system. Change from Baseline to end of study (EOS) in safety laboratory, vital signs and physical examination will be summarized in appropriate tables.
The safety and tolerability, as evaluated by medicinal use during study, following single, twice-daily (BID) and repeated BID ascending doses of Apo-Si-K170A-C76 following IN in healthy participants. | 5 days
  Concomitant medications entered into the database will be coded using the public World Health Organization (WHO) Drug Reference List, which employs the Anatomical Therapeutic Chemical classification system.
Number of participants with abnormal laboratory tests | 5 days
  Blood and urine samples were collected for the assessment of laboratory tests. Number of participants with abnormal laboratory test parameters (i.e. outside normal parameter tests results from baseline to EOS) are presented.
Number of participants with physical examination | 5 days
  Physical examination was performed extensively and focally throughout the study duration, from baseline to EOS. Number of participants with abnormal physical examination are presented.
Number of participants with abnormal vital signs | 5 days
  Vital signs were measured in a semi-supine position after five minutes of rest and included temperature, systolic blood pressure (SBP), diastolic blood pressure (DBP) , heart rate, respiratory rate. Number of participants with abnormality in any vital signs from baseline to EOS are presented.

SECONDARY OUTCOMES:
Systemic exposure be determined by measuring serum concentrations (ng/ml) of Apo-Si-K170A-C76 obtained in each cohort, at specific time points. | 5 days
  Bioanalytical analysis of the concentration of the active drug in serum samples

CONTACTS AND LOCATIONS:
Overall Officials: Hagit Grimberg, PhD, Study Director — Interna Therapeutics Ltd.; Yoseph Caraco, MD, Principal Investigator — HCRC Ein Karem, Israel
Locations (1):
- HCRC Ein Karem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Translating the vision of macromolecule therapeutics into a druggable reality — https://interna.bio/

DOCUMENTS (2):
  • Study Protocol (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT07095049/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT07095049/SAP_001.pdf